CLINICAL TRIAL: NCT00485576
Title: A Randomized, Double Blind, Placebo-Controlled, Crossover Study to Evaluate the Safety and Efficacy of Eculizumab in Subjects With Mild Allergic Asthma.
Brief Title: Safety and Efficacy Study of Eculizumab in Patients With Mild Allergic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Alexion Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C07-002
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: Allergic Asthma
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: eculizumab — eculizumab 600 mg or matching placebo iv infusion.

SUMMARY:
This study is to designed to test the role of complement in the late asthmatic response to allergen challenge in mild asthma, as an indicator of the possible role of complement in the broader asthmatic population.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with stable, mild, allergic asthma;
* history of episodic wheeze and shortness of breath;
* sexually active women of childbearing potential must use contraceptive during the entire duration of study;
* willing and able to give informed consent;
* positive methacholine challenge;
* positive skin prick test to common aeroallergens;
* positive allergen-induced early and late phase bronchoconstrictor response
* FEV1 at least 70% of predicted value;
* PC20 at baseline that is within 1 doubling dose of that measured during screening

Exclusion:

* active bacterial infection;
* respiratory tract infection or worsening of asthma within 28 days
* use of inhaled or topical steroids within 28 days or use of systemic corticosteroids within 90 days;
* use of cromoglycate, nedocromil, leukotriene receptor antagonists and inhibitors of 5-lipoxygenase within 14 days;
* use of antihistamines, immunosuppressives, or any medications that interact with eculizumab;
* use of theophylline-containing agents (any type), long-acting beta 2-agonists (salmeterol, formoterol) or long-acting anticholinergics within 14 days;
* use of NSAIDs prior to spirometry;
* use of tobacco products currently or within the previous 12 months; or smoking history > 10 pack-years;
* lung disease other than mild allergic asthma;
* patients with LAR who have not been vaccinated against Neisseria meningitidis;
* hepatitis B or HIV infection;
* parasitic infection;
* participation in any other investigational drug trial;
* pregnant or breast feeding women, or intending to conceive during the course of trial;
* known hypersensitivity to the treatment drug or any of its excipients;
* history of illicit drug use or alcohol abuse within previous year;
* any clinically significant abnormality on screening lab test results;
* abnormal chest X-ray;
* chronic use of any other medication for treatment of allergic lung disease other than short-acting beta2-agonists or ipratropium bromide;
* any medical condition that might interfere with the subject's participation in the study or confound the assessment of the subject;
* unwilling or inability to comply with the study protocol for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Allergen-induced late asthmatic response as measured by the AUC of FEV1 from 3 to 7 hours post-allergen challenge | 7 hours

SECONDARY OUTCOMES:
At 24 hours post-allergen challenge; treatment comparison of allergen-induced changes from baseline in sputum eosinophils and metachromatic cells | 72 hours
Allergen-induced airway responsiveness 24 hours post-allergen challenge as primary interest; 72 hour assessment timepoint will be supportive | 72 hours
Maximum % decrease in FEV1 from 3 to 7 hours post-allergen challenge | 7 hours
% decrease of FEV1 at 24 hours post-allergen challenge | 24 hours
AUC and maximum % fall of FEV1 from 0-3 hours post-allergen challenge | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Henk-Andre Kroon, MD, Study Director — Alexion Pharmaceuticals, Inc.
Locations (2):
- Canada (2):
  - McMaster University, Hamilton, Ontario
  - Hospital Laval, Ste-Foy, Quebec